CLINICAL TRIAL: NCT04427852
Title: Nutrition, Vision, and Cognition in Sport Study: Beef
Acronym: IONSport:Beef
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Steven E.Riechman, PhD, MPH, Associate Professor, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M1803347
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Change; Nutrient Deficiency; Nutritional Anemia; Visual Spatial Processing; Diet, Healthy; Diet; Deficiency; Dietary Deficiency; Dietary B12 Deficiency; Dietary Zinc Deficiency; Dietary Vitamin B12 Deficiency Anemia; Dietary Deficiency of Selenium and Vitamin E
MeSH Terms: conditions — Spatial Processing; Malnutrition

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either one serving of beef or a macronutrient equivalent "veggie patty" per day for 30 days.
Masking Description: note on masking: The title of the study presented to participants is "IONsport: Women and Protein" and the funding source is withheld to mask from participants our underlying hypothesis. It is open label in the sense that they know what they are eating.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 30 day Beef consumption (Experimental): One serving of beef is consumed each day for 30 days.
  Interventions: Dietary Supplement: 30 day Daily consumption of 1 serving of beef
- 30 day Veggie Patty consumption (Placebo Comparator): One serving (1 patty) of a vegetable based protein source is consumed each day for 30 days. The weight of the food, total calories, grams of protein, and total fat are the same as the beef serving.
  Interventions: Dietary Supplement: 30 day Daily consumption of 1 serving of the vegatable protein source

INTERVENTIONS:
Dietary Supplement: 30 day Daily consumption of 1 serving of beef — Beef patty will replace one of the participants protein servings each day for 30 days. Each serving is 114 grams of 90% lean ground sirloin given to participants as an uncooked frozen patty.
  Arms: 30 day Beef consumption
Dietary Supplement: 30 day Daily consumption of 1 serving of the vegatable protein source — Veggie patty will replace one of the participants protein servings each day for 30 days. No beef will be consumed during this period. The veggie patty is commercially available Morningstar veggie burger and is given to participants in commercial packaging as a frozen precooked patty.
  Arms: 30 day Veggie Patty consumption

SUMMARY:
The purpose of this study is to determine whether a 30 day beef intervention can improve peak cognitive performance in young, normally menstruating adult women. The control group will consume a daily portion of macronutrient equivalent vegetable source of protein.

DETAILED DESCRIPTION:
The purpose of the Nutrition, Vision, and Cognition in Health Sport: Beef (IONSport-Beef) study is to conduct a randomized controlled trial to evaluate beef as a nutritional intervention to optimize visual cognitive training performance in generally healthy, normally menstruating women. Female subjects of reproductive age (18-40) will be randomly placed in one of two dietary treatment groups: one serving of beef per day for 30 days or a non-meat protein replacement control. Cognitive performance will be measured in 15 training sessions over 10 days using the sophisticated NeuroTracker™ CORE (NT) 3-Dimensional (3D) software program. It is hypothesized that women consuming 1 serving of beef per day for 30 days will have the highest plasma levels of the beef rich nutrients and demonstrate the highest visual cognitive performance and improvement as compared to the no beef control.

ELIGIBILITY:
Inclusion Criteria:

1. 18-40 year old female
2. Eumenorrheic

Exclusion Criteria:

1. Neuroactive medications such as Ritalin, Adderall, antidepressants etc
2. Dietary supplements
3. Iron intake above 15mg/day
4. Protein intake above 1.5 g/kg/day
5. More than 1 mild concussion lifetime or 1 mild concussion within the last 12 months
6. History of affective disorder
7. Visual impairments uncorrected by glasses
8. Amenorrhea or dysmenorrhea
9. Currently being treated for anemia
10. >3 servings of beef per week
11. <20 BMI or BMI >35
12. Consume >100mg caffeine/day (>1 cup of coffee or soda)
13. <1 hour/week physical activity, >4 hours/week vigorous activity
14. Depression score >18 (Beck Depression Inventory)
15. <20 Kcal/kg/day

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Biological female, normally menstruating
Enrollment: 80 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Mean NeuroTracker Speed Threshold over 300 trials | 15 sessions (300 trials) over 10 days at the end of the nutritional intervention
  Cognitive Performance on the Neurotracker 3D software program that includes 20 trials in each session. Particpants will track 4 of 8 balls with increasing speed if successful and slower if unsuccessful.The speed threshold is optimized performance for that session. Across the 15 sessions, mean speed threshold is defined as the average speed threshold for the 15 sessions.
Maximal NeuroTracker Speed Threshold over 300 trials | 15 sessions (300 trials) over 10 days at the end of the nutritional intervention
  Cognitive Performance on the Neurotracker 3D software program that includes 20 trials in each session. Particpants will track 4 of 8 balls with increasing speed if successful and slower if unsuccessful. The speed threshold is optimized performance for that session. Across the 15 sessions, maximal speed threshold is defined as the highest speed threshold.
Change in NeuroTracker Speed Threshold over 300 trials | 15 sessions (300 trials) over 10 days at the end of the nutritional intervention
  Cognitive Performance on the Neurotracker 3D software program that includes 20 trials in each session. Particpants will track 4 of 8 balls with increasing speed if successful and slower if unsuccessful. The speed threshold is optimized performance for that session. Across the 15 sessions, change in speed threshold is defined as the difference between the mean of the first three sessions and the mean of the last three sessions.

SECONDARY OUTCOMES:
Blood Markers of anemia | Day 1 and Day 30 of the intervention
  blood levels of B12, iron, CBCs, ferritin, hepcidin

CONTACTS AND LOCATIONS:
Overall Officials: Steve Riechman, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Will not share